CLINICAL TRIAL: NCT02394106
Title: Ofatumumab in Children With Steroid- and Calcineurin-inhibitor-resistant Nephrotic Syndrome: a Double-blind Randomized, Controlled, Superiority Trial
Brief Title: Ofatumumab in Children With Drug Resistant Idiopathic Nephrotic Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Giannina Gaslini (Other)
Responsible Party: Principal Investigator, Gian Marco Ghiggeri MD, PhD, MD, director of Nephrology, Dialysis and Transplantation Unit, Istituto Giannina Gaslini
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OFA1
Record Dates: First submitted 2015-03-06; First posted 2015-03-20 (Estimated); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Nephrotic Syndrome
MeSH Terms: conditions — Nephrotic Syndrome | interventions — ofatumumab; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ofatumumab (Experimental): * Drug Name: Ofatumumab
  * Why: Anti-body/antigen interaction results in cell apoptosis and reduced CD20 positive cell related activities
  * Procedures: methylprednisolone 2 mg/kg infused in 30' IV diluted in 100 ml of normal saline (NaCl 0,9%); oral paracetamol 15 mg/kg ; cetirizine 0,4 mg/kg IV infused slowly in 5 ml of normal saline (NaCl 0,9%) prior to Ofatumumab infusion to reduce common reactions
  * Who provides: registered nurse
  * How: Ofatumumab IV at 12 ml/hour in the first 30'. Thereafter, the infusion rate can be doubled every 30 minutes up to a maximum of 200 ml/hour.
  * Where: in Hospital
  * When and how much: once; diluted in 1000 ml of normal saline
  * Tailoring: 1500 mg/1.73m2
  * How well: expert nurse would assist administration
  Interventions: Drug: Ofatumumab
- Placebo (Placebo Comparator): * Drug Name: Normal Saline (NaCl 0,9%)
  * Why: standard therapy could not be used as comparator for Ofatumumab, given its toxicity and lack of effectiveness. Moreover, although Rituximab, a chimeric monoclonal anti-CD20 antibody, is increasingly being used as a steroid-sparing treatment option for children with certain forms of INS (those that respond to and are dependent of steroids), this drug does not work in DR-INS and could not be used as a comparator.
  * Materials and Procedures: The placebo arm will receive the same infusion as the Ofatumumab Arm with the exception of the Ofatumumab.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ofatumumab — Ofatumumab 1500 mg/1.73m2 administered once, diluted in 1000 ml of normal saline
  Other Names: Arzerra
  Arms: Ofatumumab
Other: Placebo — Normal saline, 1000 ml, administered once
  Other Names: Normal saline
  Arms: Placebo

SUMMARY:
Double-blind, two-parallel-arm, placebo-controlled randomized clinical trial testing the superiority of Ofatumumab versus placebo in the treatment of children with DR-INS. Participants will be stratified according to eGFR at enrollment.

Eligible participants will enter a 3-months run-in period, during which instructions on urine collection and dipstick readings will be carefully reviewed, compliance assessed and any immunosuppressive therapies withdrawn according to the following schemes:

* prednisone will be tapered off by 0.3 mg/kg per week until complete withdrawal;
* calcineurin inhibitors and mofetile mycophenolate will be decreased by 50% and withdrawn after 2 additional weeks In order to minimize the risk of complications of uncontrolled INS a treatment with ACE-inhibitor at 6 mg/m2 will be maintained or started in all patients.

After run-in period, children will be randomized to the intervention arm (Ofatumumab) or comparator arm (placebo). Randomization will be stratified by eGFR at randomization: ≥90 and <90 ml/min/1.73 m2.

All patients will be followed up to 12 months and they will leave the study at time of relapse.

Relapse will be defined as uPCR ≥2000 mg/g (≥200 mg/mmol) or ≥ 3+ protein on urine dipstick for 3 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* Drug resistance: it signifies lack of antiproteinuric effect of a double therapy based on steroid plus CNI or mofetil mycophenolate (MMF). Steroid resistance is defined by failure to achieve complete remission after 6 weeks with prednisone 60 mg/m2. CNI (cyclosporine/tacrolimus) resistance is defined by failure to achieve complete remission within 6 months after the plasma concentration of cyclosporine (started at dosage of 4 mg/kg/day) or tacrolimus (started at dosage of 0,1 mg/kg/day) reached effective plasma concentrations. Mofetil Mycophenolate resistance is defined by failure to achieve complete remission after at least 6 months of treatment with 1200mg/mq/day.
* Parents'/guardian's written informed consent, and child's assent given before any study-related procedure not part of the subject's normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to his or her future medical care.
* Age between 2 and 18 years
* Histological pattern of minimal change disease, mesangial proliferation with IgM deposits or focal segmental glomerulosclerosis

Exclusion Criteria:

* Positivity to autoimmunity tests (ANA, dsDNA, ANCA).
* Reduction of C3 levels.
* eGFR < 30 ml/min/1.73 m2 valuated according to revised Bedside Schwartz Formula for patients between 2 and 17 years and with CKD-EPI Creatinine 2009 Equation for 18 years old patients.
* Hystological pattern characterized by elements suggestive for congenital disease: diffuse mesangial sclerosis without IgM deposits, cystic-like tubular dilatation, mitochondrial abnormalities evident on electron microscopy, IF suggestive for congenital collagen 4 disease.
* Histological pattern not suitable with INS in the pediatric age (membranous glomerulonephritis, lupus nephritis, diffuse and/or localized vasculitis, amyloidosis)
* Homozygous or heterozygous mutations of podocitary genes, commonly involved in the etiology of INS (NPHS1, NPHS2, NPHS3, NPHS6, WT1, COQ2, COQ6, MYO1E, SMARCAL1, LAMB2, SCARB2, CD2AP, TRPC6, ACTN4, INF2, LMX1B, MYH9 )
* Pregnancy
* Neoplasm
* Infections: Previous or actual HBV (with HBeAb positivity) or HCV

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2015-07; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Complete or partial disease remission | 6 months from randomization
  Complete remission in defined by urinary protein/creatinine ratio (uPCR) <200 mg/g (<20mg/mmol) for 3 consecutive days. Partial remission is defined as proteinuria reduction of 50% or greater from the presenting value and absolute uPCR between 200 and 2000 mg/g. for 3 consecutive days (according to KDIGO Clinical Practice Guideline for Glomerulonephritis)

SECONDARY OUTCOMES:
Complete or partial disease remission | 12 months from randomization;
  Complete remission in defined by urinary protein/creatinine ratio (uPCR) <200 mg/g (<20mg/mmol) for 3 consecutive days. Partial remission is defined as proteinuria reduction of 50% or greater from the presenting value and absolute uPCR between 200 and 2000 mg/g. for 3 consecutive days (according to KDIGO Clinical Practice Guideline for Glomerulonephritis)
Adverse events | At 1, 3, 6, 9 and 12 months after drug/placebo infusion, during protocol visits
  Measurement of frequency and severity of adverse events due to drug infusion
Abnormal laboratory values | At 1, 3, 6, 9 and 12 months after drug/placebo infusion, during protocol visits
  Record of abnormal values in biochemical tests and hematology assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Gianmarco Ghiggeri, MD, Principal Investigator — Istituto Giannina Gaslini
Locations (1):
- IRCCS Istituto Giannina Gaslini, Genoa, Italy/GE, Italy

REFERENCES:
- [Background] Basu B. Ofatumumab for rituximab-resistant nephrotic syndrome. N Engl J Med. 2014 Mar 27;370(13):1268-70. doi: 10.1056/NEJMc1308488. No abstract available. PMID 24670185
- [Background] Robak T. Ofatumumab, a human monoclonal antibody for lymphoid malignancies and autoimmune disorders. Curr Opin Mol Ther. 2008 Jun;10(3):294-309. PMID 18535937
- [Background] Magnasco A, Ravani P, Edefonti A, Murer L, Ghio L, Belingheri M, Benetti E, Murtas C, Messina G, Massella L, Porcellini MG, Montagna M, Regazzi M, Scolari F, Ghiggeri GM. Rituximab in children with resistant idiopathic nephrotic syndrome. J Am Soc Nephrol. 2012 Jun;23(6):1117-24. doi: 10.1681/ASN.2011080775. Epub 2012 May 10. PMID 22581994
- [Background] Ravani P, Magnasco A, Edefonti A, Murer L, Rossi R, Ghio L, Benetti E, Scozzola F, Pasini A, Dallera N, Sica F, Belingheri M, Scolari F, Ghiggeri GM. Short-term effects of rituximab in children with steroid- and calcineurin-dependent nephrotic syndrome: a randomized controlled trial. Clin J Am Soc Nephrol. 2011 Jun;6(6):1308-15. doi: 10.2215/CJN.09421010. Epub 2011 May 12. PMID 21566104
- [Background] Ravani P, Rossi R, Bonanni A, Quinn RR, Sica F, Bodria M, Pasini A, Montini G, Edefonti A, Belingheri M, De Giovanni D, Barbano G, Degl'Innocenti L, Scolari F, Murer L, Reiser J, Fornoni A, Ghiggeri GM. Rituximab in Children with Steroid-Dependent Nephrotic Syndrome: A Multicenter, Open-Label, Noninferiority, Randomized Controlled Trial. J Am Soc Nephrol. 2015 Sep;26(9):2259-66. doi: 10.1681/ASN.2014080799. Epub 2015 Jan 15. PMID 25592855
- [Background] McEnery PT, Strife CF. Nephrotic syndrome in childhood. Management and treatment in patients with minimal change disease, mesangial proliferation, or focal glomerulosclerosis. Pediatr Clin North Am. 1982 Aug;29(4):875-94. No abstract available. PMID 7050865
- [Background] Ghiggeri GM, Catarsi P, Scolari F, Caridi G, Bertelli R, Carrea A, Sanna-Cherchi S, Emma F, Allegri L, Cancarini G, Rizzoni GF, Perfumo F. Cyclosporine in patients with steroid-resistant nephrotic syndrome: an open-label, nonrandomized, retrospective study. Clin Ther. 2004 Sep;26(9):1411-8. doi: 10.1016/j.clinthera.2004.09.012. PMID 15531003
- [Background] Radhakrishnan J, Cattran DC. The KDIGO practice guideline on glomerulonephritis: reading between the (guide)lines--application to the individual patient. Kidney Int. 2012 Oct;82(8):840-56. doi: 10.1038/ki.2012.280. Epub 2012 Aug 15. PMID 22895519
- [Background] Caridi G, Bertelli R, Di Duca M, Dagnino M, Emma F, Onetti Muda A, Scolari F, Miglietti N, Mazzucco G, Murer L, Carrea A, Massella L, Rizzoni G, Perfumo F, Ghiggeri GM. Broadening the spectrum of diseases related to podocin mutations. J Am Soc Nephrol. 2003 May;14(5):1278-86. doi: 10.1097/01.asn.0000060578.79050.e0. PMID 12707396
- [Derived] Liu ID, Willis NS, Craig JC, Hodson EM. Interventions for idiopathic steroid-resistant nephrotic syndrome in children. Cochrane Database Syst Rev. 2025 May 8;5(5):CD003594. doi: 10.1002/14651858.CD003594.pub7. PMID 40337980
- [Derived] Ravani P, Pisani I, Bodria M, Caridi G, Degl'Innocenti ML, Ghiggeri GM. Low-dose ofatumumab for multidrug-resistant nephrotic syndrome in children: a randomized placebo-controlled trial. Pediatr Nephrol. 2020 Jun;35(6):997-1003. doi: 10.1007/s00467-020-04481-y. Epub 2020 Jan 28. PMID 31993781